CLINICAL TRIAL: NCT03116373
Title: Impact of Tracheal Tube Fixing Site on Its Mobility During Head Mobilization
Acronym: Fix-IOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 29BRC17.0025
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Intubation, Intratracheal
Keywords: Posture; Physiology; Head; Intubation; Intratracheal methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- maxilla fixing then mandible fixing (Active Comparator): The tracheal tube is first fixed on the maxilla. After the measures of the outcomes, its site of fixation is changed for the mandible for the outcome measurement in the second site of fixation.
  Interventions: Other: mandible fixation; Other: Maxilla fixation
- mandible fixing then maxilla fixing (Active Comparator): The tracheal tube is first fixed on the mandible. After the measures of the outcomes, its site of fixation is changed for the maxilla for the outcome measurement in the second site of fixation.
  Interventions: Other: mandible fixation; Other: Maxilla fixation

INTERVENTIONS:
Other: mandible fixation — Intubation device will be fixed on mandible
Other: Maxilla fixation — Intubation device will be fixed on maxilla

SUMMARY:
This study evaluate the secondary shifting of the tracheal tube when the head is moved under general anaesthesia. Two sites of fixation (the maxilla and the mandible) are tested in a prospective, double blind, randomized and crossover designed study.

The study test the hypothesis that taping the tracheal tube on the mandible better prevents a secondary tube move.

DETAILED DESCRIPTION:
Tracheal intubation is the only technique to ensure airway protection, meaning preventing aspiration, and providing mechanical ventilation during general anesthesia (GA). This is an extremely frequent procedure. After intubation, the head of the patient is often moved as the patient is positioned for the surgical procedure (ENT, thoracic and abdominal surgeries, lateral or prone positioning…). This may even happen several times during the same procedure. It is well demonstrated that these head movements are responsible for secondary shifting of the tube (1-9). This can cause accidental extubation or selective bronchial intubation.

The anesthesiologist secures the tube with tape to prevent secondary displacement of the tracheal tube. The two most common sites to tape the tube on patient's face are the maxilla, because it is a fixed spot on the face, and the mandible, because its mobility coming from the temporomandibular joint may allow a better interlock with the larynx.

There is no study and no recommendation about the best site of tape. Both techniques are commonly used, depending on the anesthesiologist's preference.

Investigators designed a, controlled study in Brest university hospital to compare two groups by cross-over intervention (one group "maxilla fixing then mandible fixing" and one group "mandible fixing then maxilla fixing").

The population is composed of adult patients undergoing bronchoscopy or endobronchial ultrasound under GA and after tracheal intubation. The bronchoscope allows a permanent control of the tracheal tube's position, and the possibility of shifting it without compromising patient security, which is not possible in other daily surgical procedure.

Statisticien estimate that the total number of patients to include is 36. In order to avoid a sequence effect, the order of the fixing technique will be randomized. Every patient will be its own control as there is a cross over-design.

The main outcome is the maximal amplitude of the tracheal tube shifting when the head is bended on the chest and extended in the back, controlled by bronchoscopy with each fixing technique.

The anesthesiologist investigator will use the first fixing site according to the patient's randomization group. Then, he will display an opaque cover around the tracheal tube, so that the operator, who will measure the tube displacements, will stay blind. As the intervention is performed under GA, the patient will also be blind. The same procedure will be performed after the second fixing site is used, before the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Bronchoscopy or endobronchial ultrasound
* General anaesthesia
* Tracheal intubation

Exclusion Criteria:

* Patient incapable of consenting or with a legal guardian or declining participation
* Forbidden or impaired cervical mobility (less than 80°)
* Mouth opening less than 35 mm
* Moustache or Beard

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Maximal amplitude of the tracheal tube shifting | 2 minutes
  The main outcome is the maximal amplitude of the tracheal tube shifting when the head is bended on the chest and extended in the back, controlled by bronchoscopy with each fixing technique.

SECONDARY OUTCOMES:
Movement of the tracheal tube from the neutral position | 2 minutes
  For each fixation site (maxillary or mandibular), the tracheal tube displacement from the neutral position is measured when the head is bended on the chest and when it is extended in the back.

CONTACTS AND LOCATIONS:
Locations (1):
- Brest University Hospital, Brest, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Conrardy PA, Goodman LR, Lainge F, Singer MM. Alteration of endotracheal tube position. Flexion and extension of the neck. Crit Care Med. 1976 Jan-Feb;4(1):8-12. doi: 10.1097/00003246-197601000-00002. No abstract available. PMID 1253616
- [Result] Yap SJ, Morris RW, Pybus DA. Alterations in endotracheal tube position during general anaesthesia. Anaesth Intensive Care. 1994 Oct;22(5):586-8. doi: 10.1177/0310057X9402200515. PMID 7818064
- [Result] Hartrey R, Kestin IG. Movement of oral and nasal tracheal tubes as a result of changes in head and neck position. Anaesthesia. 1995 Aug;50(8):682-7. doi: 10.1111/j.1365-2044.1995.tb06093.x. PMID 7645696
- [Result] Sugiyama K, Yokoyama K. Displacement of the endotracheal tube caused by change of head position in pediatric anesthesia: evaluation by fiberoptic bronchoscopy. Anesth Analg. 1996 Feb;82(2):251-3. doi: 10.1097/00000539-199602000-00006. PMID 8561322
- [Result] Rost JR, Frush DP, Auten RL. Effect of neck position on endotracheal tube location in low birth weight infants. Pediatr Pulmonol. 1999 Mar;27(3):199-202. doi: 10.1002/(sici)1099-0496(199903)27:33.0.co;2-o. PMID 10213259
- [Result] Olufolabi AJ, Charlton GA, Spargo PM. Effect of head posture on tracheal tube position in children. Anaesthesia. 2004 Nov;59(11):1069-72. doi: 10.1111/j.1365-2044.2004.03963.x. PMID 15479313
- [Result] Weiss M, Knirsch W, Kretschmar O, Dullenkopf A, Tomaske M, Balmer C, Stutz K, Gerber AC, Berger F. Tracheal tube-tip displacement in children during head-neck movement--a radiological assessment. Br J Anaesth. 2006 Apr;96(4):486-91. doi: 10.1093/bja/ael014. Epub 2006 Feb 7. PMID 16464981
- [Result] Jordi Ritz EM, Von Ungern-Sternberg BS, Keller K, Frei FJ, Erb TO. The impact of head position on the cuff and tube tip position of preformed oral tracheal tubes in young children. Anaesthesia. 2008 Jun;63(6):604-9. doi: 10.1111/j.1365-2044.2008.05440.x. PMID 18477271
- [Result] Kim JT, Kim HJ, Ahn W, Kim HS, Bahk JH, Lee SC, Kim CS, Kim SD. Head rotation, flexion, and extension alter endotracheal tube position in adults and children. Can J Anaesth. 2009 Oct;56(10):751-6. doi: 10.1007/s12630-009-9158-y. Epub 2009 Jul 29. PMID 19639372